CLINICAL TRIAL: NCT00842179
Title: Femoral Access Site Groin Complication Rates After 2517 Groin Punctures Undergoing Vascular Closure by Either Manual Compression or the Perclose Vascular Closure Device
Brief Title: Groin Complications Post Percutaneous Coronary Intervention Using Either Manual Compression or PERCLOSE Device
Status: Completed | Type: Observational
Sponsor: Clinyx, LLC (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Holly Taylor, Clinyx
Other Study IDs: CL-003
Record Dates: First submitted 2009-02-06; First posted 2009-02-12 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Vascular Closure
Keywords: Perclose

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Manual Closure: Patients who received vascular closure with manual compression after percutaneous coronary intervention (PCI)
- Perclose Device: Patients who received vascular closure with the Perclose VCD after percutaneous coronary intervention (PCI)

SUMMARY:
The objective of this study is to compare groin complication rates in low and high risk patients post percutaneous coronary intervention (PCI) closed by either a 6 French Perclose vascular closure device (VCD) or manual compression.

DETAILED DESCRIPTION:
It is commonly accepted that that there exists a learning curve in performing successful groin closure with Vascular Closure Devices (VCD). Manual compression continues to be 'standard of care' at most institutions for closure of 5 - 8 French femoral arteriotomies, as previous studies evaluating the safety and efficacy of vascular closure devices have failed to show a statistically significant decrease in groin complication rates when compared to manual compression. Importantly, no studies to date have been performed to specifically assess the potential decrease in vascular complication rates by highly experienced VCD operators, when their safety results are compared to manual compression. This retrospective, multi-center study will demonstrate a lower vascular complication rate in PCI patients post deployment of a 6 Fr Perclose VCD by a single, experienced operator, when compared to manual compression in two comparable, high volume, hospital cardiac catheterization laboratories.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received vascular closure with the Perclose device post PCI at Baptist Miami Hospital
* Patients who received vascular closure by manual compression at Tampa General Hospital

Exclusion Criteria:

* Patients less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who require vascular closure post percutaneous coronary intervention
Sampling Method: Probability Sample
Enrollment: 2517 (Actual)
Dates: Start 2008-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
major vascular complications | 0-30 days (during Index hospitalization)

SECONDARY OUTCOMES:
Minor vascular complications | 0-30 days (during index hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Roberts, MD, Principal Investigator — Baptist Health South Florida
Locations (1):
- Baptist Hospital of Miami, Miami, Florida, United States